CLINICAL TRIAL: NCT01780558
Title: A Randomized Controlled Study:the Different Outcomes Between Natural Cycle and Hormon Replacement Cycle in FET
Brief Title: A Study:the Different Outcomes Between Natural Cycle and Hormone Replacement Cycle in FET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qingxue Zhang, professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-design-FET
Record Dates: First submitted 2013-01-24; First posted 2013-01-31 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Infertility
Keywords: endometrium preparation protocols; frozen-thawed embryo transfer; natural cycles; hormone replacement therapy cycles; randomized controlled trial
MeSH Terms: conditions — Infertility | interventions — Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group NC-A (Other): Patients with regular cycles undergoing FET in reproductive medicine renter of Sun Yat-sen Memorial Hospital will be recruited, who should not be elder than 40 and had more than 3 frozen embryos.They will be randomized to receive the natural cycles.
  Interventions: Other: natural cycles
- group HRT-B (Other): Patients with regular cycles undergoing FET in reproductive medicine renter of Sun Yat-sen Memorial Hospitalwill be recruited , who should not be elder than 40 and had more than 3 frozen embryos will be randomized to receive the estradiol and progesterone replacement therapy cycles.
  Interventions: Drug: estradiol and progesterone

INTERVENTIONS:
Other: natural cycles — the ovulation is monitored spontaneously or induced by HCG when the dominant follicle is larger than 18mm without LH surge. Transfer of thawed embryos will be performed 4 days after LH surge/HCG administration or 3 days after ovulation is observed.
  Other Names: spontaneous ovulation cycles
  Arms: group NC-A
Drug: estradiol and progesterone — oral estradiol, 2 mg, once daily, is introduced on cycle day 3 with an increasing doses protocol. If the endometrial thickness is greater than 7mm, progesterone 40-60 mg in oil will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later.
  Other Names: Estradiol Valerate; Progynova; corpus luteum hormone; luteal hormone
  Arms: group HRT-B

SUMMARY:
There are three main cycle regimens used for endometrial preparation for frozen embryo transfer（FET）: natural cycles (NC) with/without ovulation triggering, hormone replacement therapy cycles (HRT) in which the endometrium is artificially prepared by estrogen and progesterone hormones with/without a gonadotrophin releasing hormone agonist (GnRH-a) down regulation, and ovulation induced cycles (OI) in which follicular development is supported with increasing doses of gonadotrophin hormones and ovulation is induced. At present, there is still no sufficient evidence that which kind of FET cycle regimen to plan more advantage. The purpose of this study was to compare the pregnancy outcome of NC-FET to that of HRT-FET in women with regular cycles.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial. Patients with regular cycles undergoing FET in reproductive medicine renter of Sun Yat-sen Memorial Hospital will be recruited，who should not be elder than 40 and had more than 3 frozen embryos. They will be randomized to receive either the NC-FET cycle (group NC-A) or the HRT-FET cycle (group HRT-B). In group NC-A, the ovulation is monitored spontaneously or induced by human chorionic gonadotropin(HCG) when the dominant follicle is larger than 18mm without luteinizing hormone surge(LH). Transfer of thawed embryos will be performed 4 days after LH /HCG administration or 3 days after ovulation is observed. In group HRT-B, oral estradiol, 2 mg, once daily, is introduced on cycle day 3 with an increasing doses protocol. If the endometrial thickness is greater than 7mm, progesterone 40-60 mg in oil will be administered via intramuscular injection. Transfer of thawed embryos will be performed 3 days later. This study was approved by the reproductive medicine ethics committee of Sun Yet-sen Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age forty years old or less
* Has regulation Menstruation (cycle 24-35 days) or previous data suggest that normal ovulation
* Frozen embryos number more than three

Exclusion Criteria:

* Has Chocolate cyst or adenomyosis of uterus
* Clear hydrosalpinx
* Uterine scar or intrauterine adhesion and endometrial thickness <7mm before ovulation
* recur thick endometrium（<7mm）
* repeated implantation failure（≥3 times）
* Cancel the cycle because of having no dominant follicle in the NC+FET before or the growth of endometrium not good in the HRT+FET before

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Live-birth rate | Live-birth after FET

SECONDARY OUTCOMES:
pregnancy rate | 2 weeks after Embryo transplantation
  2 weeks after Embryo transplantation, people go urine HCG and blood HCG test，positive as pregnancy
clinical pregnancy rate | 5 weeks after Embryo transplantation
  5 weeks after Embryo transplantation,people go Vaginal B ultrasonic，being saw the gestation sac as clinical pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Zhang qingxue, doctor, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China